CLINICAL TRIAL: NCT03473964
Title: Adrenocorticotrophic Hormone (ACTH) for the Treatment of Sarcoid Uveitis
Brief Title: (ACTH) for the Treatment of Sarcoid Uveitis
Acronym: ACTH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: John Huang, MD (Other)
Responsible Party: Sponsor-Investigator, John Huang, MD, MD ophthalmologist, New England Retina Associates
Organization: New England Retina Associates (Other)
Other Study IDs: 1169914
Record Dates: First submitted 2018-01-31; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Sarcoid Uveitis
MeSH Terms: interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment: The study intervention is the observation of study subjects who have received H.P. Acthar® Gel (adrenocorticotrophic hormone), 40 units twice weekly injections in patients who have sarcoid uveitis and to assess it's effectiveness by measuring changes the degree of aqueous and vitreous inflammatory cells present, the degree of aqueous flare, and changes in visual acuity, macular thickness, intraocular pressure and quality of life measures assessed by using the National Eye Institute Visual Function Questionnaires (VFQ-25)
  Interventions: Drug: H.P. Acthar gel

INTERVENTIONS:
Drug: H.P. Acthar gel — H.P. Acthar gel:
  Injection 40 mg twice weekly
  Other Names: adrenocorticotrophic hormone

SUMMARY:
Sarcoidosis is a multisystem granulomatous disease that can affect nearly any organ in the body. While most commonly affecting the lungs, vision threatening eye involvement occurs in approximately 25% of patients with sarcoid. Eye involvement may lead to a chronic, sight-threatening uveitis which may result in cataract, glaucoma, and macular edema. The treatment of sarcoid uveitis involves the use of topical and systemic corticosteroids or potent immunosuppressive agents (medications that suppress the body's immune system) both of which can cause severe long-term side effects. The adverse effects of steroids may be avoided by treatment with the use as H.P. Acthar® Gel. The effectiveness of H.P. Acthar® Gel in the treatment of sarcoid uveitis and patient quality of live have not been previously examined. These issues, will be explored in this research.

DETAILED DESCRIPTION:
The Investigator seeks to determine the efficacy of H.P. Acthar® Gel (40 units twice weekly injection) of on disease activity and severity in patients with sarcoid uveitis. The retrospective study will evaluate a series of quantitative outcome measures:

The degree of aqueous and vitreous inflammatory cells as graded by the criteria established by the Standardization of Uveitis Nomenclature (SUN) criteria at intervals of 0 weeks, 3 weeks, 6 weeks, 12 weeks and 24 weeks.

The degree of aqueous flare as graded by the criteria established by the Standardization of Uveitis Nomenclature (SUN) criteria at intervals of 0 weeks, 4 weeks,12 weeks and 24 weeks.

Best Corrected Visual Acuity at intervals of 0 weeks, 4 weeks, 12 weeks and 24 weeks.

Central Macular Thickness at intervals of 0 weeks, 4 weeks, 12 weeks and 24 weeks as measured by Optical Coherence Tomography (OCT).

Intraocular pressure at intervals of 0 weeks, 4 weeks, 12 weeks and 24 weeks as measured by applanation tonometry

Quality of life assessment using National Eye Institute Visual Function Questionnaire (VFQ-25)

The Investigator expects to retrospectively review the charts of 10 sarcoid associated uveitis patients treated with Acthar® Gel over a period of 1 year.

ELIGIBILITY:
Inclusion Criteria:

Presence of Sarcoid Uveitis as determined by

* clinical exam
* fluorescence angiography
* optical coherence tomography

Exclusion Criteria:

* Presence of long acting intraocular depots
* Women of childbearing age not using contraceptives

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with sarcoid uveitis with disease activity, as determined by clinical exam, fluorescein angiography and optical coherence tomography.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Degree of aqueous and vitreous inflammatory cells-change is being assessed | 0 weeks, 4 weeks, 12 weeks and 24 weeks.
  Degree of aqueous and vitreous inflammatory cells as graded by the criteria established by the Standardization of Uveitis Nomenclature (SUN)

SECONDARY OUTCOMES:
Degree of aqueous flare- change is being assessed | 0 weeks, 4 weeks 12 weeks and 24 weeks
  Degree of aqueous flare as graded by the criteria established by Standardization of Uveitis Nomenclature (SUN)
Visual acuity- change is being assessed | 0 weeks, 4 weeks, 12 weeks and 24 weeks
  Testing and evaluation of best corrected visual acuity using Luxvision trial frames and Precision Vision ETDRS charts R,1 and 2
Central macular thickness- change is being assessed | 0 weeks, 4 weeks, 12 weeks and 24 weeks
  Central macular thickness as measured by Spectralis Optical Coherence Tomography (OCT)
Intraocular pressure | 0 weeks, 4 weeks, 12 weeks and 24 weeks
  Intraocular pressure as measured by applanation tonometry
Quality of life assessment- change is being assessed | 0 weeks, 4 weeks, 12 weeks and 24 weeks
  Quality of life assessment using the National Eye Institute Visual Function Questionnaire (VFQ-25). The VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single item general health rating question. The scoring ranges in scores from 1-6, 1 being activity presents no difficulty and 6 being can no longer perform this activity due to vision. The VFQ-25 generates the following vision-targeted subscales : global vision rating (1), difficulty with near vision activities (3), difficulty with distance vision activities (3), limitations in social functioning due to vision (2), role limitations due to vision(2), dependency on others due to vision (3), mental health symptoms due to vision (4), driving difficulties (3), limitations with peripheral (1) and color vision (I), and ocular pain (2).

CONTACTS AND LOCATIONS:
Overall Officials: John J Huang, MD, Principal Investigator — New England Retina Associates
Locations (1):
- New England Retina Associates, Hamden, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided